CLINICAL TRIAL: NCT05850364
Title: A Multi-country, Multi-center, Open-labelled, Randomized, Controlled, Extended Phase Ⅲ Clinical Trial to Evaluate the Immunogenicity and Tolerability of Sabin Strain Inactivated Poliovirus Vaccine Administered With or Without Routine Infant Vaccines
Brief Title: A Multi-center, Open-labelled, Randomized, Controlled, Extended Phase Ⅲ Clinical Trial of sIPV Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-sIPV-4001
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Poliomyelitis; Polio
Keywords: Polio vaccines; Poliomyelitis Vaccine; Inactivated polio vaccine; Sabin Inactivated Poliovirus Vaccine (sIPV)
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group C1 (Experimental): Co-administration of sIPV and routine infant vaccines at 6,10,14 weeks old (N=360)
  Interventions: Biological: Sabin Strain Inactivated Poliovirus Vaccine
- group C2 (Experimental): Co-administration of sIPV and routine infant vaccines at 6, 10,14 weeks old
  Interventions: Biological: Sabin Strain Inactivated Poliovirus Vaccine
- group S1 (Experimental): Administration of sIPV at 6,10,14 weeks old; Administration of routine infant vaccines at 8,12,16 weeks old
  Interventions: Biological: Sabin Strain Inactivated Poliovirus Vaccine
- group S2 (Experimental): Administration of routine infant vaccines at 6,10,14 weeks old; Administration of sIPV at 8,12,16 weeks old
  Interventions: Biological: Sabin Strain Inactivated Poliovirus Vaccine

INTERVENTIONS:
Biological: Sabin Strain Inactivated Poliovirus Vaccine — Totally 1440 healthy infants of 6 weeks old (42-47 days) are planned to be enrolled, and then randomized in a 1:1:1:1 ratio into four groups, i.e., co-administration group 1 (group C1), co-administration group 2 (group C2), staggered administration group 1 (group S1) and staggered administration group 2 (group S2). Participants in group C1 and C2 will receive sIPV at 6,10, 14 weeks old, administered concomitantly with routine infant vaccine (may include DTP-HepB-Hib vaccine, PCV10 or rotavirus vaccine in accordance with the local routine vaccination schedule). Participants in group S1 will receive sIPV at 6,10,14 weeks old, and receive routine infant vaccines at 8,12,16 weeks old. Participant s in group S2 will receive routine infant vaccines at 6,10,14 weeks old, and receive sIPV at 8,12, 16 weeks old.

SUMMARY:
This study is designed to study the immunogenicity and safety of sIPV co-administered with other routine infant vaccines. According to the national immunization schedule of Bangladesh and Pakistan, sIPV was administered concomitantly with PCV10, DTP-HeB-Hib and other vaccines at 6, 10 and 14 weeks old. Thus, this study set up the concomitant vaccination schedule according to the real practice in study area. The primary hypothesis of this study is the seroconversion rate of polio vaccination when administered concomitantly with routine vaccines, is non-inferior to that when administered alone; the secondary hypothesis of this study is the seropositivity rate of diphtheria, tetanus, and pertussis when routine vaccines are administered concomitantly with sIPV, is non-inferior to that administered without sIPV.

DETAILED DESCRIPTION:
This is a multi-country, multi-center, open-labelled, randomized, controlled, extended phase Ⅲ clinical trial. Totally 1440 healthy infants of 6 weeks old (42-47 days) are planned to be enrolled, and then randomized in a 1:1:1:1 ratio into four groups, i.e., co-administration group 1 (group C1), co-administration group 2 (group C2), staggered administration group 1 (group S1) and staggered administration group 2 (group S2). Participants in group C1 and C2 will receive sIPV at 6,10, 14 weeks of age, administered concomitantly with routine infant vaccine (may include DTP-HepB-Hib vaccine, PCV10 or rotavirus vaccine in accordance with the local routine vaccination schedule). Participants in group S1 will receive sIPV at 6,10,14 weeks of age, and receive routine infant vaccines at 8,12,16 weeks of age. Participants in group S2 will receive routine infant vaccines at 6,10,14 weeks of age, and receive sIPV at 8,12, 16 weeks old.

For all the Participants, the immediate reactions within 30 minutes after each dose of vaccination will be observed on site. Guardians of participants will utilize the diary card to record solicited adverse events from the time of vaccination for 7 days post-vaccination of each dose. From the time of the first vaccination and 28 days post-vaccination of the last dose, unsolicited adverse events and any SAEs will be required to recorded in the diary card.

About 3 ml venous blood will be collected before the first vaccination and 28 days (+7) days after the last vaccination of sIPV or routine vaccines. Antibodies level will be determined using the collected sera for immunogenicity evaluation. Group C1 and S1 will be compared in terms of immunogenicity against polio; Group C2 and S2 will be compared in terms of immunogenicity against diphtheria, Tetanus, Pertussis, Hepatitis B, Hib and Pneumococcal.

ELIGIBILITY:
Inclusion Criteria:

1) Infants of 6 weeks old (42-47 days); 2) For whom a parent/legal guardian has given written informed consent after the study has been explained; 3) Be able to provide the vaccination records after birth; 4) Negative results in SARS-CoV-2 rapid antigen testing, within 24 hours before enrollment; 5) The participant's mother was tested negative for HIV, Syphilis, Hepatitis A, Hepatitis B infection during or before (during pregnancy) her child's enrollment to this study (the test result should be provided, and that obtained during pregnancy is acceptable).

-

Exclusion Criteria:

1) History of polio vaccination (except the OPV at birth); 2) Prior vaccination with routine infant vaccines against Diphtheria, Tetanus, Pertussis, Haemophilus influenzae type b (Hib), Pneumococcal or rotavirus; 3) History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component; 4) Infants with premature labor (delivery before week 37 of gestation) and low body weight (birth body weight is <2500 g); 5) Infants with difficult labor at birth, asphyxiation rescue and history of nervous system injury; 6) Congenital malformation or development disorder, genetic defect, severe malnutrition, etc.; 7) Autoimmune disease or immunodeficiency/immunosuppression; 8) Patients with serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia, or neurological disorders); 9) Abnormal coagulation functions (such as coagulation factor deficiency, blood coagulation disease and blood platelet disorders) or obvious bruise or blood coagulation disorders diagnosed by the doctors; 10) Those who have received immunosuppressant therapy, cytotoxic drug therapy and inhaled corticosteroid therapy (excluding the corticosteroid aerosol therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis); 11) The volunteer has received blood products before inoculation of the trial vaccine; 12) The volunteer has received other study drugs within 30 days before inoculation of the trial vaccine; 13) The volunteer has received live attenuated vaccines within 14 days before inoculation of the trial vaccine; 14) The volunteer has received subunit or inactivated vaccines within 7 days before inoculation of the trial vaccine; 15) Various acute diseases or acute exacerbation of chronic diseases within recent 7 days; 16) Significant acute disease or chronic infection within the previous 7 days or axillary temperature equal and more than 37.3℃ prior to vaccination in the present study; 17) The volunteer has any other factors which are unsuitable for participation in the clinical trial as judged by the investigators.

-

Ages: 42 Days to 47 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1442 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the non-inferiority of immune response to polio vaccination, when administered concomitantly with routine vaccines | 28 days
  Seroconversion rates of neutralizing antibody against polioviruses of three serotypes, at 28 days after three doses of vaccinationadministered concomitantly with routine vaccines
To evaluate the safety in terms of ARs (Vaccine-related AEs） | 7 days
  Incidence of adverse reactions within 7 days after each dose of vaccination Incidence of adverse reactions within 7 days after each dose of vaccination

SECONDARY OUTCOMES:
To evaluate non-inferiority of immune response to diphtheria and tetanus antigens, when routine vaccines are administered concomitantly with sIPV | 28 days
  Seropositivity rate of IgG antibodies against diphtheria and tetanus, at 28 days after vaccination
To evaluate non-inferiority of immune response to acellular pertussis antigens, when routine vaccines are administered concomitantly with sIPV | 28 days
  Seropositivity rate of IgG antibodies against pertussis toxin (PT), Filamentous hemagglutinin (FHA), Pertactin (PRN), at 28 days after vaccination
To evaluate the immunogenicity against hepatitis B and Hib, when routine vaccines are administered concomitantly with sIPV | 28 days
  Sero-protection rate of IgG antibodies against hepatitis B and Hib, at 28 days after vaccination and GMC of IgG antibodies against hepatitis B and Hib, at 28 days after vaccination
To evaluate the immunogenicity against pneumococcal, when routine vaccines are administered concomitantly with sIPV | 28 days
  Sero-protection rate of IgG antibodies against pneumococcal, at 28 days after vaccination and GMC of IgG antibodies against pneumococcal, at 28 days after vaccination
To evaluate other immunogenicity of sIPV, when administered concomitantly with routine vaccines | 28 days
  GMT of neutralizing antibodies against polioviruses of three serotypes, at 28 days after three doses of vaccination
To evaluate other immunogenicity against diphtheria, tetanus, acellular pertussis antigens | 28 days
  GMC of IgG antibodies against diphtheria, tetanus, acellular pertussis antigens, at 28 days after vaccination
To evaluate the safety in terms of SAEs | 14 months
  Incidence of SAEs throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Wasif A Khan, Dr., Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (3):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh
- Pakistan (2):
  - Central Hospital, Gujranwala
  - The Aga Khan University, Karachi

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05850364/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT05850364/SAP_001.pdf